CLINICAL TRIAL: NCT01811862
Title: Acupuncture for Symptom Control in Hematopoietic Stem Cell Transplantation Patients: A Pilot Study
Brief Title: Acupuncture for Symptom Control in Hematopoietic Stem Cell Transplantation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-038
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Multiple Myeloma
Keywords: Acupuncture; Hematopoietic stem cell transplantation (HSCT); 13-038
MeSH Terms: conditions — Multiple Myeloma | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Acupuncture (Experimental): Acupuncture treatment once daily inpatient for 5 consecutive days starting at on the day after chemotherapy plus usual pre- and post-transplantation care.
  Interventions: Procedure: Acupuncture
- Sham acupuncture (Sham Comparator): Sham acupuncture once daily inpatient for 5 consecutive days starting at on the day after chemotherapy plus usual pre- and post-transplantation care.
  Interventions: Procedure: Sham acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Patients with multiple myeloma undergoing conditioning myeloablative chemotherapy followed by autologous hematopoietic stem cell transplantation. Patients will be randomized to acupuncture or sham acupuncture. Acupuncture treatment will be delivered once daily starting on Day -1 (Day -2 is the day chemotherapy starts). Acupuncture will continue for 5 days, or, when the patient's absolute neutrophil count drops below 200/microliter or platelet count drops below 20,000/microliter, whichever is sooner. Sham acupuncture will be delivered on the same schedule. Regardless of group assignment, every patient will receive the same usual prevention and treatment regimen for nausea, vomiting, anxiety, insomnia and fatigue that other patients who are undergoing conditioning chemotherapy in preparation for HSCT will receive in the Transplant Service.
  Arms: Acupuncture
Procedure: Sham acupuncture — Patients with multiple myeloma undergoing conditioning myeloablative chemotherapy followed by autologous hematopoietic stem cell transplantation. Patients will be randomized to acupuncture or sham acupuncture. Acupuncture treatment will be delivered once daily starting on Day -1 (Day -2 is the day chemotherapy starts)Acupuncture will continue for 5 days, or, when the patient's absolute neutrophil count drops below 200/microliter or platelet count drops below 20,000/microliter, whichever is sooner. Sham acupuncture will be delivered on the same schedule. Regardless of group assignment, every patient will receive the same usual prevention and treatment regimen for nausea, vomiting, anxiety, insomnia and fatigue that other patients who are undergoing conditioning chemotherapy in preparation for HSCT will receive in the Transplant Service.
  Arms: Sham acupuncture

SUMMARY:
This is a prospective randomized controlled trial to obtain preliminary data for the design of a future definitive efficacy study. A randomized controlled trial is needed because comparison to historical data would be biased. The investigators will use sham acupuncture as the control to account for effect from attention from and interaction with the therapist.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or above (those age below 21 are usually treated in the Pediatric Transplant Service)
* Diagnosis of multiple myeloma
* Scheduled to receive conditioning chemotherapy followed by upfront or salvage autologous peripheral blood hematopoietic stem cell transplantation

Exclusion Criteria:

* Absolute neutrophil count less than 200/microliter
* Platelet count less than 20,000/microliter
* Acupuncture treatment in the preceding 4 weeks prior to Day 1

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-03; Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
whether acupuncture reduces common symptoms | 2 years
  In patients undergoing chemotherapy prior to hematopoietic stem cell transplantation. The primary endpoint is the area-under-curve (AUC) for MDASI total score from Day -2 to Day 5. MDASI scores are assessed daily by having the patient fill out the questionnaire. Severity is assessed for the 13 core MDASI symptom items (pain, fatigue, nausea, disturbed sleep, distress etc..) AUC for MDASI total score from Day -2 to Day 5 will be compared between the acupuncture group and the sham acupuncture group.

SECONDARY OUTCOMES:
to assess the effect size for each symptom | 2 years
  Effect size for each symptom will be calculated descriptively. To determine whether baseline characteristics predict response to acupuncture, each will be added as an interaction term to the primary model. The following predictors will be explored: inpatient vs outpatient treatment, upfront vs. salvage transplantation, age, baseline MDASI score, pro-inflammatory cytokine levels, and use of symptom control medications (yes / no).

CONTACTS AND LOCATIONS:
Overall Officials: Gary Deng, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] El Iskandarani S, Sun L, Li SQ, Pereira G, Giralt S, Deng G. Acupuncture improves certain aspects of sleep in hematopoietic stem cell transplantation patients: a secondary analysis of a randomized controlled trial. Acupunct Med. 2023 Dec;41(6):319-326. doi: 10.1177/09645284231181403. Epub 2023 Jul 6. PMID 37409464
- [Derived] Deng G. Acupuncture As a Potential Opioid-Sparing Pain Management Intervention for Patients Undergoing Cancer Treatment. Med Acupunct. 2020 Dec 1;32(6):394-395. doi: 10.1089/acu.2020.1494. Epub 2020 Dec 16. PMID 33362896
- [Derived] Deng G, Giralt S, Chung DJ, Landau H, Siman J, Li QS, Lapen K, Mao JJ. Reduction of Opioid Use by Acupuncture in Patients Undergoing Hematopoietic Stem Cell Transplantation: Secondary Analysis of a Randomized, Sham-Controlled Trial. Pain Med. 2020 Mar 1;21(3):636-642. doi: 10.1093/pm/pnz190. PMID 31498394
- [Derived] Deng G, Giralt S, Chung DJ, Landau H, Siman J, Search B, Coleton M, Vertosick E, Shapiro N, Chien C, Wang XS, Cassileth B, Mao JJ. Acupuncture for reduction of symptom burden in multiple myeloma patients undergoing autologous hematopoietic stem cell transplantation: a randomized sham-controlled trial. Support Care Cancer. 2018 Feb;26(2):657-665. doi: 10.1007/s00520-017-3881-7. Epub 2017 Sep 17. PMID 28920142
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/